CLINICAL TRIAL: NCT02421471
Title: Post-Marketing Surveillance to Evaluate the Safety and Efficacy of Picato® Gel
Brief Title: PMS to Evaluate the Safety and Efficacy of Picato® Gel
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PICATO-1130
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2018-01

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; topical treatment; ingenol mebutate
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ingenol mebutate treatment cohort: Patients who are prescribed ingenol mebutate gel for the first time by investigator's medical judgment.
  Interventions: Drug: Ingenol mebutate 0.015 percent or 0.05 percent gel

INTERVENTIONS:
Drug: Ingenol mebutate 0.015 percent or 0.05 percent gel — Topical treatment with ingenol mebutate gel 0.015 percent or 0.05 percent gel of skin areas affected by AK
  Other Names: Picato®

SUMMARY:
This study is a mandatory post launch observational study in South Korea of 3.000 patients receiving treatment for the first time with a new medicinal product, ingenol mebutate gel (Picato®), approved for topical treatment of actinic keratosis.

Each patient is observed for 8 weeks after treatment completion.

DETAILED DESCRIPTION:
Picato® (ingenol mebutate) gel is a new topical therapy for Actinic Keratosis (AK) in adults which was approved by the Korean Ministry of Food and Drug Safety (MFDS) in December 2013. For AK in face or scalp the 0.015 percent gel is approved to be applied once a day for 3 consecutive days, and for AK in trunk or extremities the 0.05 percent gel is approved to be applied once a day for 2 consecutive days.

The re-examination period for Picato® runs from December 2013 to December 2019, during which at least 3,000 patients who are prescribed ingenol mebutate gel for the first time by investigator's medical judgment must be documented in a standard Post Marketing Surveillance (PMS) study.

Each patient is to be observed for 8 weeks following application of ingenol mebutate gel. If a patient is unable to visit the PMS site, the investigator may contact the patient by phone to assess the safety.

ELIGIBILITY:
Inclusion Criteria:

Adult patient with AK First time treatment with ingenol mebutate 0.015 or 0.05 percent gel

Exclusion Criteria:

* Children and adolescents

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients with AK in involved PMS sites treated for the first time with ingenol mebutate 0.015 or 0.05 percent gel.
Sampling Method: Non-Probability Sample
Enrollment: 1324 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 8 weeks after treatment completion
  According to Korean definition and classification, covering serious as well as non-serious Adverse Events, related as well as non-related to ingenol mebutate treatment
Overall improvement | 8 weeks after treatment completion
  Graded by investigator on a 3-point scale ('improved', 'no change', 'worsened'), based on number of AK lesions in treated area compared to baseline

SECONDARY OUTCOMES:
Complete clearance rate - Change in AK lesions count: Percentage (%) change in the total number of AK lesions compared to baseline* | 8 weeks after treatment
  Proportion of patients with no clinically visible AK lesions in treated area
Partial clearance rate | 8 weeks after treatment
  Proportion of patients with 75% or greater reduction in the number of AK lesions in treated area compared to baseline
Change in AK lesion count | 8 weeks after treatment
  Percentage change in the total number of AK lesions in treated area compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sun Choi, B.Sc., Study Director — LEO Pharma Limited, Korea
Locations (1):
- Department of Dermatology, Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No